CLINICAL TRIAL: NCT03441035
Title: Albumin Mass Balance in Liver Transplantation, an Open Prospective Cohort Study
Brief Title: Albumin Mass Balance in Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ake Norberg (Other)
Responsible Party: Sponsor-Investigator, Ake Norberg, Associate professor, Senior Consultant, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Other Study IDs: K2017-4774; 4-3344/2017 (Other: Karolinska Institutet)
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Liver Transplant; Complications; Fluid Overload
MeSH Terms: conditions — Edema | interventions — Anesthesia, General; Surgical Procedures, Operative; Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma for determination of P-albumin, Plasma for determination of markers of inflammation and endothelial dysfunction or injury (such as interleukine 6, syndecan, heparin-binding protein), X-albumin to be determined in urine, succion bottles, drains, and any albumin containing intravenous infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adults, uncomplicated: Adults undergoing liver transplantation. Mass balance of albumin will be undertaken by sampling of albumin in plasma and in all fluids that is infused or lost from the body to keep track of albumin and hemoglobin changes until postoperative day 7. B-Hb is taken routinely and not study specific samples. Plasma for ELISAs is taken at 2-3 time points.
  Interventions: Other: General anesthesia and surgery (liver transplantation)
- Adults, complicated: Adults undergoing liver transplantation. Mass balance of albumin will be undertaken by sampling of albumin in plasma and in all fluids that is infused or lost from the body to keep track of albumin and hemoglobin changes until hospital discharge or postoperative day 21. B-Hb is taken routinely and not study specific samples. Plasma for ELISAs is taken at 2-3 time points. A infusion of deuterium labeled phenylalanine will be given in the ICU at 1-3 occasions to determine the synthesis rate of albumin.
  Interventions: Other: General anesthesia and surgery (liver transplantation)
- Children: Children undergoing liver transplantation. Mass balance of albumin will be undertaken by sampling of albumin in in all fluids that is infused or lost from the body to keep track of albumin and hemoglobin changes until postoperative day 7. P-albumin and B-Hb is only taken routinely and not study specific samples. Plasma for ELISAs is taken at 2-3 time points.
  Interventions: Other: General anesthesia and surgery (liver transplantation)

INTERVENTIONS:
Other: General anesthesia and surgery (liver transplantation) — The effects of general anesthesia and surgery under the hospital routine of albumin administration during and after liver transplantation is studied with the mass balance of albumin method.

SUMMARY:
This clinical observational cohort study assess the loss of albumin from blood circulation during and after liver transplantation by mass balance of albumin. The overall assumption of this method is that if albumin is more diluted than hemoglobin, it must have left the plasma, presumably into the interstitial space. Predictors of albumin leakage will be assessed, including biomarkers of inflammation and of endothelial damage and dysfunction. The sub cohorts children and patients with complications, defined as prolonged postoperative treatment in the intensive care unit, respectively, will be focused in separate publications.

DETAILED DESCRIPTION:
Background Capillary leakage has been recognized to be associated with surgery and inflammation [Fleck 1985]. In liver transplantation considerable amounts of exogenous albumin is administered to support circulatory stability and a post operative plasma albumin concentration of 25 g/L to facilitate interpretation of immuno suppressive drug concentrations. However, the long term effects of exogenous albumin is not well characterized in the literature, and extravasation might promote edema formation and impair wound healing. In previous studies we have demonstrated the ability of the albumin mass balance method to identify leakage of albumin in major abdominal surgery [Norberg 2016].

In a pilot study in patients undergoing liver transplantation (n=11) we found a net leakage of albumin from plasma of 37 ± 17 g at end of surgery and 48 ± 33 g at postoperative day 3.

The primary aim of the new study is to find if this net leakage is still there at postoperative day 7. We are also looking into predictors of positive albumin shift from plasma including markers of inflammation and endothelial injury or dysfunction. Focus will also be put on the subgroup of children during and after liver transplantation. Finally a subgroup of patients in need of prolonged ICU stay after liver transplantation will be investigated to see the prolonged effects of our present routines, and these patients ability to synthetize albumin.

All patients undergoing liver transplantation at Karolinska University Hospital are eligible.

Recruitment will be made in advance as soon as patients are put on the transplant waiting list. In adults, at the day of surgery, blood samples will be taken repeatedly for estimation of plasma albumin. In all patients we will keep track of any gains or losses of albumin or hemoglobin in suction bottles, drains, exogenous blood products, exogenous albumin etc. This sampling will proceed during the study period that will end at hospital discharge or not later than post-operative day 21. Adult patients that are still in the ICU on postoperative day 3 will be subjected to a measurement of albumin synthesis rate by the flooding method [Ballmer 1993]. All subjects, even children, will have blood sampled for ELISAs of markers of inflammation and endothelial injury or dysfunction.

Total study specific blood sampling will be limited to 100 mL in adults and 6 mL in children.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing liver transplantation are eligible

Exclusion Criteria:

No consent Unability to understand the study information (language or consciousness)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing liver transplantation at our unit (approximately 85 patients per year) will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative perioperative shift of albumin | Post-operative day 7 after liver transplantation
  By mass balance of albumin (i.e keeping track of all gains and losses of albumin and compare these to hemoglobin) it is possible to estimate the loss of albumin from plasma that is not explained by losses in bleeding or drains.

SECONDARY OUTCOMES:
Predictors of cumulative perioperative shift of albumin | from pre-operative risk assessment until post-operative day 7
  anthropometric and laboratory values including markers of inflammation and endothelial injury or dysfunction will be analyzed by regression analysis to cumulative perioperative shift of albumin
Predictors of prolonged need for ICU stay | from pre-operative risk assessment until post-operative day 21
  anthropometric and laboratory values including markers of inflammation and endothelial injury or dysfunction will be analyzed by regression analysis to Patients in need or not in need of prolonged ICU treatment
Albumin synthesis rate | postoperative days 3-21 after liver transplantation
  By deuterium labeled phenylalanine it is possible to assess albumin synthesis rate by the "flooding technique"
Cumulative perioperative shift of albumin in children | during and after liver transplantation until postoperative day 21
  By mass balance of albumin (i.e keeping track of all gains and losses of albumin and compare these to hemoglobin) it is possible to estimate the loss of albumin from plasma that is not explained by losses in bleeding or drains.

CONTACTS AND LOCATIONS:
Overall Officials: Åke Norberg, Ass Prof, Principal Investigator — Perioperative Medicine and Intensive Care, Karolinska University Hospital Huddinge
Locations (1):
- Karolinska University Hospital, Huddinge, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleck A, Raines G, Hawker F, Trotter J, Wallace PI, Ledingham IM, Calman KC. Increased vascular permeability: a major cause of hypoalbuminaemia in disease and injury. Lancet. 1985 Apr 6;1(8432):781-4. doi: 10.1016/s0140-6736(85)91447-3. PMID 2858667
- [Background] Norberg A, Rooyackers O, Segersvard R, Wernerman J. Leakage of albumin in major abdominal surgery. Crit Care. 2016 Apr 26;20(1):113. doi: 10.1186/s13054-016-1283-8. PMID 27117323
- [Background] Ballmer PE, McNurlan MA, Milne E, Heys SD, Buchan V, Calder AG, Garlick PJ. Measurement of albumin synthesis in humans: a new approach employing stable isotopes. Am J Physiol. 1990 Dec;259(6 Pt 1):E797-803. doi: 10.1152/ajpendo.1990.259.6.E797. PMID 2260648

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT03441035/Prot_SAP_000.pdf